CLINICAL TRIAL: NCT01242683
Title: Case-Management & Environmental Support to Sustain Weight Loss & Reduce CHD Risk
Brief Title: Vivamos Activos Fair Oaks Program for Weight Loss in Low Income Latinos
Acronym: VAFO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: San Mateo Medical Center (Other); El Concilio of San Mateo County (Unknown); Palo Alto Medical Foundation (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Randall Stafford, Randall S. Stafford MD, PhD, Professor of Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SU-10112010-7069; R01HL089448 (NIH)
Record Dates: First submitted 2010-11-15; First posted 2010-11-17 (Estimated); Last update posted 2014-06-02 (Estimated); Status verified 2014-05

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Case-Management for Behavior Change (Experimental): Individual and group sessions devoted to behavioral strategies to facilitate weight loss conducted by a health educator. 12 month of intensive intervention followed by 12 months of maintenance intervention.
  Interventions: Behavioral: Vivamos Activos Fair Oaks Program
- Case-Management plus Home Visits (Experimental): Community health worker lifestyle support for weight loss strategies conducted in participants' homes and neighborhood. Also, receive individual and group sessions devoted to behavioral strategies to facilitate weight loss conducted by a health educator. 12 month of intensive intervention followed by 12 months of maintenance intervention.
  Interventions: Behavioral: Vivamos Activos Fair Oaks Program
- Usual Primary Care (Placebo Comparator): Continuation of usual primary care managed by the participants' usual physician or nurse practitioner source of care.
  Interventions: Behavioral: Vivamos Activos Fair Oaks Program

INTERVENTIONS:
Behavioral: Vivamos Activos Fair Oaks Program — Comparison of Case-management vs. Case-management plus Home Visits vs. Usual Primary Care.
  Case-management: Five 60 minute individual and 15 90 minute group sessions devoted to behavioral strategies to facilitate weight loss conducted by a health educator.
  Home-visits: Seven home visits provided by a community health worker to provide life-style/environmental support for behavior change to facilitate weight loss.
  Usual primary care: Usual care provided at health center that is available to participants in all three study arms.
  Other Names: Modified and Tailored Diabetes Prevention Program Protocol

SUMMARY:
Physician-based primary care has thus far failed to address the obesity epidemic. In this randomized clinical trial of 200 obese patients with heart disease risk factors, the investigators will evaluate the impact of nurse and dietitian case management on weight loss and weight maintenance, as an adjunct to physician care. In addition, the investigators will test the incremental benefit of an environmental support strategy using community health workers to help patients navigate their home and neighborhood environments to achieve weight loss. The innovative intervention model developed and evaluated in this project has the potential to provide a blueprint for successful primary care-based obesity services

DETAILED DESCRIPTION:
Obesity is an epidemic in the U.S., with a third of adults obese. Obesity exerts enormous impact on the nation's health and economy largely through its effect on coronary heart disease (CHD) risk factors: 3 in 4 obese Americans have at least one CHD risk factor reversible through weight loss. Working within acute care-centered systems, most clinicians are unsuccessful in helping their patients lose weight or prevent weight gain. A promising and well-studied approach is integrated care delivered by nurse and dietitian case managers (CMs). Nonetheless, clinical prevention services (including CM) may be less effective if provided in isolation from patients' living environments that so often reinforce caloric excess and physical inactivity.

This application leverages our extensive expertise in developing and disseminating effective CM programs (Heart to Heart, R01 HL070781). We will implement an obesity-focused CM program that focuses on established behavioral weight loss and maintenance strategies and evidence-based CHD prevention targets. We also will test the additional benefit of structured "environmental support" (ES) carried out by community health workers that will bridge the gap between the clinic and patients' homes and neighborhood. Our Specific Aims are to:

1. Implement innovative, primary care-based CM and CM+ES interventions in a randomized clinical trial. We will conduct this trial at a San Mateo Medical Center (SMMC) health center serving an ethnically diverse, low-income population. We will randomize 200 obese adults with at least one obesity-related CHD risk factor over 18 months to usual primary care (40 patients), CM alone (80), or CM+ES (80). Intervention patients in will receive an intensive weight loss and CHD risk intervention for 12 months, followed by 12 months of maintenance intervention.
2. Determine the effectiveness and cost-effectiveness of the CM and CM+ES for improving BMI and CHD risk factors, relative to usual care and each other. Our PRIMARY HYPOTHESIS is that patients managed through CM+ES will experience greater reductions in BMI over 24-months than those in CM.
3. Transition the favored intervention to a sustainable program, supported by the County, as well as explore opportunities for broader dissemination to other County and non-County systems. A business case for dissemination based on our findings will be critical in seeking this investment.

This project will develop and test two novel models of care design to support sustained weight loss. Given the failure of current mechanisms to address obesity and elevated CHD risk, these models have the potential to provide a blueprint for primary care-based obesity services that can reduce this nation's burden of obesity, especially for low-income populations.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older;
2. Body mass between 30 and 55 kg/m2
3. One or more CHD risk factors: Systolic blood pressure between 130 and 200 mmHg; Diastolic blood pressure between 80 and 105 mmHg; Total cholesterol > 180 mg/dL; LDL cholesterol > 120 mg/dL; HDL Cholesterol < 40 mg/dL; Triglycerides > 150 mg/dL; HbA1c between 6.0 and 11.5%; Fasting plasma glucose between 95 and 400 mg/dL; Diagnosis of Type 2 diabetes
4. Residing in catchment area of the Fair Oaks Adult Clinic and receiving primary care at Fair Oaks Adult Clinic.

Exclusion Criteria:

1. Inability to speak Spanish;
2. Unwilling to attempt weight loss;
3. Significant medical co-morbidities, including uncontrolled metabolic disorders (e.g., thyroid, diabetes, renal, liver), unstable heart disease, advanced heart failure, and ongoing substance abuse;
4. On greater than 10 prescription medications;
5. Psychiatric disorders requiring antipsychotics or multiple medications;
6. Body weight change > 25 lbs. in the preceding 3 months;
7. Pregnant, planning to become pregnant, or lactating less than six months;
8. Family household member already enrolled in the study;
9. Intends to or is enrolled in a study that would limit full participation in VAFO;
10. Participants who are unwilling to have home visits by study staff;
11. Resident of a long term care facility;
12. Plans to move during the study period (24 months post-randomization);
13. Investigator discretion for clinical safety or adherence reasons (e.g., unstable housing, chronic pain).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2008-05; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
body mass index | 24 months

SECONDARY OUTCOMES:
blood lipid measurements | 24 months
Fasting blood glucose | 24 months
triglycerides | 24 months
Hemoglobin A1c | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Randall S. Stafford MD, PhD, Principal Investigator — Stanford University
Locations (4):
- United States (4):
  - Palo Alto Medical Foundation Research Institute, Palo Alto, California
  - San Mateo Medical Center, Fair Oaks Adult Clinic, Redwood City, California
  - El Concilio of San Mateo, San Mateo, California
  - Stanford University School of Medicine, Stanford, California

REFERENCES:
- [Background] Drieling RL, Ma J, Stafford RS. Evaluating clinic and community-based lifestyle interventions for obesity reduction in a low-income Latino neighborhood: Vivamos Activos Fair Oaks Program. BMC Public Health. 2011 Feb 14;11:98. doi: 10.1186/1471-2458-11-98. PMID 21320331
- [Derived] Drieling RL, Goldman Rosas L, Ma J, Stafford RS. Community resource utilization, psychosocial health, and sociodemographic factors associated with diet and physical activity among low-income obese Latino immigrants. J Acad Nutr Diet. 2014 Feb;114(2):257-265. doi: 10.1016/j.jand.2013.07.025. Epub 2013 Oct 8. PMID 24119533